CLINICAL TRIAL: NCT07036016
Title: Interstitial Pneumonitis Associated With EGFR-TKI and Combined With PD-1/PD-L1: A Retrospective Observational Study In Patients With Non-Small Cell Lung Cancer
Brief Title: Interstitial Pneumonitis Associated With EGFR-TKI and Combined With PD-1/PD-L1
Status: Completed | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: WHUH_2025_06
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- EGFR-TKI
  Interventions: Drug: EGFR-TKI
- PD-1/PD-L1
  Interventions: Drug: PD-1/PD-L1 inhibitor
- EGFR-TKI combined with PD-1/PD-L1
  Interventions: Drug: EGFR-TKI combined with PD-1/PD-L1

INTERVENTIONS:
Drug: EGFR-TKI — epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKIs)-including gefitinib, erlotinib, afatinib, and osimertinib
  Groups: EGFR-TKI
Drug: PD-1/PD-L1 inhibitor — ICIs such as nivolumab, pembrolizumab, and atezolizumab-targeting the programmed cell death 1 (PD-1) or its ligand (PD-L1)
  Groups: PD-1/PD-L1
Drug: EGFR-TKI combined with PD-1/PD-L1 — epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKIs)-including gefitinib, erlotinib, afatinib, and osimertinib combined with ICIs such as nivolumab, pembrolizumab, and atezolizumab-targeting the programmed cell death 1 (PD-1) or its ligand (PD-L1)
  Groups: EGFR-TKI combined with PD-1/PD-L1

SUMMARY:
Importance:

EGFR tyrosine kinase inhibitors (EGFR-TKIs) and PD-1/PD-L1 immune checkpoint inhibitors are widely used in the treatment of non-small cell lung cancer (NSCLC). However, the safety profile of their combination-particularly the risk of interstitial pneumonitis (IP)-remains unclear.

Objective:

To evaluate the incidence and risk of interstitial pneumonitis associated with EGFR-TKIs when combined with PD-1/PD-L1 inhibitors, using real-world pharmacovigilance data.

Design, Setting, and Participants:

This retrospective observational study analyzed adverse event reports from the FDA Adverse Event Reporting System (FAERS) between January 1, 2015, and December 31, 2024. A total of 67,818 NSCLC cases were included, categorized by treatment with EGFR-TKIs, PD-1/PD-L1 inhibitors, combined therapy, or the other therapies.

Exposure:

NSCLC patients receiving EGFR-TKI PD-1/PD-L1 inhibitors, combined therapy, or the other therapies were compared to those not receiving such treatment.

Main Outcome and Measures:

Incidence of reported interstitial pneumonitis and adjusted odds ratios (aORs) derived from multivariable logistic regression analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-small cell lung cancer (NSCLC).
* Received at least one EGFR-TKI (gefitinib, erlotinib, afatinib, osimertinib). Or received at least one PD-1/PD-L1 inhibitor (nivolumab, pembrolizumab, atezolizumab, durvalumab). Or received combination therapy with both EGFR-TKIs and PD-1/PD-L1 inhibitors. Or received the other therapies.
* Cases reported in the FDA Adverse Event Reporting System (FAERS) between January 1, 2015, and December 31, 2024.

Exclusion Criteria:

* Non-NSCLC Indications: Cases not related to NSCLC (e.g., other cancer types).
* Incomplete Treatment Data: Patients with missing or unclear treatment exposure information (e.g., use of unrelated therapies).
* Duplicate Reports: Duplicate adverse event reports were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 67,818 NSCLC cases were included, categorized by treatment with EGFR-TKIs, PD-1/PD-L1 inhibitors, combined therapy, or the other.
Sampling Method: Probability Sample
Enrollment: 67818 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Incidence of reported interstitial pneumonitis and adjusted odds ratios (aORs) derived from multivariable logistic regression analyses. | From January 1, 2015, and December 31, 2024

IPD SHARING:
Plan to Share IPD: Undecided